CLINICAL TRIAL: NCT06963060
Title: Xinhua Hospital A Ffiliated to Shanghai Jiaotong University School of Medicine
Brief Title: Gem+Nab-P+LEN+TIS for Advanced Unresectable BTC (GALENT-BT)
Acronym: GALENT-BT
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Wei Gong (Other)
Responsible Party: Sponsor-Investigator, Wei Gong, Xinhua Hospital A ffiliated to Shanghai Jiaotong University School of Medicine, Xinhua Hospital, Shanghai Jiao Tong University School of Medicine
Organization: Xinhua Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XHEC-C-2024-121-2
Record Dates: First submitted 2025-04-07; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Gallbladder Cancer; Cholangiocarcinoma
Keywords: advanced unresectable biliary tract malignancies
MeSH Terms: conditions — Gallbladder Neoplasms; Cholangiocarcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental): Gemcitabine ,nab-Paclitaxel,Lenvatinib and Tislelizumab
  Interventions: Drug: Gemcitabine nab-PaclitaxelLenvatinibTislelizumab

INTERVENTIONS:
Drug: Gemcitabine nab-PaclitaxelLenvatinibTislelizumab — Receive Gemcitabine (1000 mg/m² IV on Days 1 and 8) and nab-Paclitaxel (125 mg/m² IV on Days 1 and 8) every 3 weeks.
  Take Lenvatinib (4-8 mg orally daily on Days 1-21).
  Receive Tislelizumab (200 mg IV on Day 1) every 3 weeks.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of combining Gemcitabine, nab-Paclitaxel, Lenvatinib, and Tislelizumab in adults aged 18-75 years with advanced unresectable biliary tract malignancies (including gallbladder cancer, intrahepatic cholangiocarcinoma, and extrahepatic cholangiocarcinoma). The main questions it aims to answer are:

What is the objective response rate (ORR) of this quadruplet regimen as first-line therapy?

What are the secondary outcomes, including disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and safety profile?

This is a single-arm, open-label, phase II study with no comparison group.

Participants will:

Receive Gemcitabine (1000 mg/m² IV on Days 1 and 8) and nab-Paclitaxel (125 mg/m² IV on Days 1 and 8) every 3 weeks.

Take Lenvatinib (4-8 mg orally daily on Days 1-21).

Receive Tislelizumab (200 mg IV on Day 1) every 3 weeks.

Undergo 6-8 treatment cycles (adjusted for tolerability) with regular imaging, laboratory tests, and safety assessments.

Be followed for 3 years to monitor survival and long-term outcomes.

The study plans to enroll 29 participants and will be conducted at a single center over 36 months.

DETAILED DESCRIPTION:
1. Study Background Biliary tract malignancies (BTCs), including gallbladder cancer (GBC), intrahepatic cholangiocarcinoma (ICC), and extrahepatic cholangiocarcinoma (ECC), are aggressive cancers with a 5-year survival rate <5%. Current first-line systemic therapies (e.g., gemcitabine/cisplatin) yield limited efficacy (ORR <30%, median OS ~11.7 months). Preclinical and clinical evidence suggests synergistic effects of combining chemotherapy, anti-angiogenic agents, and immune checkpoint inhibitors. The GALENT-BT trial evaluates a novel quadruplet regimen-Gemcitabine + nab-Paclitaxel + Lenvatinib + Tislelizumab-to improve outcomes in advanced unresectable BTCs.
2. Study Objectives

   Primary Objective: Assess the safety and tolerability of the quadruplet regimen over 8 treatment cycles.

   Secondary Objectives:

   Evaluate objective response rate (ORR), disease control rate (DCR), progression-free survival (PFS), overall survival (OS), and surgical conversion rate.

   Monitor adverse events (AEs), serious adverse events (SAEs), and quality of life (QoL).

   Exploratory Objectives: Investigate biomarkers (e.g., PD-L1 expression, genetic mutations) and radiomic/pathologic features associated with treatment response.
3. Study Design

   Design: Prospective, single-arm, open-label, single-center, phase II trial.

   Sample Size: Two-stage enrollment:

   Stage 1 (Lead-in): 9 participants for initial safety evaluation. If ≤3/9 experience grade ≥3 AEs, proceed to Stage 2.

   Stage 2 (Expansion): 20 additional participants (total 29 evaluable patients).

   Duration: 36 months (June 2024-June 2027).
4. Study Population

   Inclusion Criteria:

   Adults aged 18-75 years with histologically confirmed, untreated, advanced unresectable BTC (GBC/ICC/ECC) or recurrent BTC (≥3 months post-adjuvant therapy).

   ECOG PS 0-1, measurable disease per RECIST 1.1, adequate organ function.

   Exclusion Criteria: Prior systemic therapy for advanced BTC, severe comorbidities, pregnancy, or intolerance to study drugs.
5. Intervention

   Regimen:

   Gemcitabine: 1000 mg/m² IV on Days 1 and 8 of each 21-day cycle.

   nab-Paclitaxel: 125 mg/m² IV on Days 1 and 8.

   Lenvatinib: 4-8 mg orally daily (weight-based dosing) on Days 1-21.

   Tislelizumab: 200 mg IV on Day 1.

   Treatment Duration: 6-8 cycles (adjustable for tolerability), followed by 3-year survival follow-up.
6. Assessments

Efficacy:

Tumor response evaluated by CT/MRI every 6 weeks using RECIST 1.1.

ORR, DCR, PFS, OS, and surgical conversion rate calculated.

Safety:

AEs/SAEs graded per CTCAE v5.0.

Laboratory monitoring (hematology, liver/renal function, thyroid panels).

QoL: Assessed via EORTC QLQ-HCC18 questionnaire at baseline, treatment cycles, and follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-75 years, regardless of gender.
2. Histologically or cytologically confirmed, untreated primary advanced unresectable biliary tract malignancies (BTC), including intrahepatic cholangiocarcinoma (ICC), extrahepatic chololiocarcinoma (ECC), and gallbladder cancer (GBC); or untreated recurrent BTC (prior adjuvant/neoadjuvant chemotherapy allowed if completed ≥3 months before recurrence, excluding regimens containing PD-1/L1 inhibitors, gemcitabine, nab-paclitaxel, or lenvatinib).
3. ECOG performance status score 0-1.
4. Expected survival ≥3 months.
5. At least one measurable target lesion per RECIST v1.1 criteria.
6. Adequate organ function:

   Hematologic: Hemoglobin ≥90 g/L; WBC ≥lower limit of normal (LLN); ANC ≥1.5×10⁹/L; platelets ≥100×10⁹/L.

   Renal: Serum creatinine ≤1.5×ULN; endogenous creatinine clearance rate ≥55 mL/min.

   Hepatic: Total bilirubin ≤1.5×ULN; ALT/AST ≤2.5×ULN (≤3×ULN for intrahepatic BTC or liver metastases; ALT/AST ≤5×ULN for liver metastases).

   Coagulation: INR ≤1.5×ULN; APTT within normal range.
7. No prior systemic therapy for advanced BTC (chemotherapy, radiotherapy, targeted therapy, immunotherapy, or hormonal therapy). Patients with post-R2 resection are eligible.
8. Negative serum/urine pregnancy test (for women of childbearing potential) and agreement to use contraception during the study and for 6 months post-treatment.
9. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Severe systemic infection or uncontrolled comorbidities (e.g., heart failure, thyroid disorders, psychiatric conditions).
2. Known hypersensitivity or intolerance to study drugs or their excipients.
3. Pregnancy, lactation, or refusal to use effective contraception.
4. Participation in other clinical trials within 30 days prior to enrollment.
5. Inability to understand or unwillingness to sign informed consent.
6. Any condition that, in the investigator's judgment, may compromise patient safety or compliance (e.g., severe concurrent illness, abnormal lab results, psychosocial factors).
7. Prior use of PD-1/L1 inhibitors, gemcitabine, nab-paclitaxel, or lenvatinib in adjuvant/neoadjuvant settings.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | At the end of Cycle 8 (each cycle is 21 days)
  The objective response rate (ORR) of this quadruplet regimen as first-line therapy

SECONDARY OUTCOMES:
Surgical Conversion Rate | At the end of Cycle 8 (each cycle is 21 days)
  The proportion of patients whose tumors become resectable after treatment and undergo curative-intent surgery (R0/R1 resection).
Disease control rate (DCR) | At the end of Cycle 8 (each cycle is 21 days)
  he proportion of patients who achieve complete response (CR), partial response (PR), or stable disease (SD)
Overall Survival (OS) | The end of the 3-year follow-up period
  Time from randomization to death from any cause
Progression-Free Survival (PFS) | At the end of disease progression or death during the 3-year follow-up period
  Time from randomization to disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Xinhua Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No